CLINICAL TRIAL: NCT06707441
Title: Which Score Best Predicts Outcomes in Chest Trauma? A Prospective Comparison of Thorax and Trauma Injury Severity Scores
Brief Title: Thorax vs. Trauma Injury Severity Scores as Outcome Predictors in Chest Trauma
Acronym: TTSS/TRISS/ER
Status: Recruiting | Type: Observational
Sponsor: Al-Nahrain University (Other)
Responsible Party: Principal Investigator, Abdul-Ilah R. Khamis, Principal Investigator, Al-Nahrain University
Other Study IDs: UNCOMIRB20241125
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Chest Trauma
Keywords: TTSS; ER; TRISS
MeSH Terms: conditions — Thoracic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this observational study is to compare the predictive utility of the Thorax Trauma Severity Score (TTSS) and the Trauma and Injury Severity Score (TRISS) in determining outcomes among patients presenting with chest trauma to the emergency room. The main questions it aims to answer are:

Does the TTSS provide a more accurate prediction of patient outcomes (e.g., mortality, ICU admission) than the TRISS? Are there specific patient subgroups where one score is more effective than the other?

Participants will:

Have their chest trauma severity assessed using both TTSS and TRISS during their emergency room admission.

Have their clinical outcomes (e.g., mortality, ICU admission, length of hospital stay) monitored throughout their hospital stay.

DETAILED DESCRIPTION:
Trauma is a significant cause of mortality and morbidity around the world. Approximately 10% of the burden of disease in adults is due to traumatic injuries. Trauma can lead to serious consequences, including disabilities, psychosocial burdens, and increased mortality among the actively working population. Cardiopulmonary arrest, unplanned admissions to intensive care units, and nosocomial infections are some complications faced by trauma patients admitted to trauma centers. The estimated mortality rate for hospitalized trauma patients is 11%. The in-hospital mortality rate for trauma patients who undergo cardiopulmonary resuscitation (CPR) is 92.7%. Trauma-related mortality and morbidity depend on injury severity, diagnostic delays, and the time taken to reach a medical facility. Timely evaluation, effective post-trauma care, and appropriate triage can significantly reduce long-term mortality and morbidity among trauma patients, with rapid assessment of trauma severity being crucial for the primary triage of multiple trauma patients.

Trauma scoring systems are essential tools in the medical field for evaluating the severity of injuries and predicting patient outcomes. Two notable scoring systems are the Thorax Trauma Severity Score (TTSS) and the Trauma and Injury Severity Score (TRISS), each serving unique purposes in assessing thoracic injuries and overall trauma severity. The TTSS was developed to provide a comprehensive assessment of thoracic injuries by incorporating both anatomical and physiological parameters. It specifically focuses on various aspects of chest trauma, including:

Age of the patient Ratio of arterial oxygen partial pressure to fractional inspired oxygen (PaO2/FiO2) Presence of pleural injuries Lung contusions Rib fractures The scoring system ranges from 0 to 25 points, where higher scores indicate more severe injuries and worse prognoses. Research has shown that a TTSS score of 7 or above is highly predictive of morbidity and mortality, achieving 100% sensitivity and 97.73% specificity for poor outcomes in isolated thoracic trauma cases. The TRISS is another critical scoring system used to evaluate overall injury severity across multiple body regions. It is based on the Injury Severity Score (ISS), which categorizes injuries according to their anatomical location using the Abbreviated Injury Scale (AIS). The ISS is calculated by taking the highest AIS scores from the three most severely injured body regions, squaring them, and summing these values.

Despite their utility, both TTSS and TRISS have limitations, especially when applied to diverse patient populations. The TTSS may not adequately account for the severity of injuries outside the thoracic region, which can significantly impact patient outcomes. For instance, a study highlighted that in patients with an Injury Severity Score (ISS) greater than 15, only 44% had a TTSS above 8, indicating that critical extra-thoracic injuries were not reflected in the TTSS scoring. Older patients or those with comorbidities may present with less obvious thoracic injuries that the TTSS fails to identify. This oversight can lead to underestimating the risk of complications or mortality, as older individuals often have a higher propensity for severe outcomes despite seemingly minor trauma. The TISS may not capture specific details related to chest trauma effectively. This limitation is crucial in regions with variable healthcare infrastructure, like Iraq, where injury mechanisms and patient demographics can differ widely. The TRISS's general approach may overlook critical factors that influence trauma severity in these populations.

This study seeks to address the specific needs of the Iraqi healthcare system by comparing the TTSS and TRISS as predictive tools for chest trauma outcomes in emergency settings. The aim is to identify which scoring system is more reliable and practical for use in Iraq, considering the unique challenges faced by emergency departments, such as high patient volumes and resource constraints. The research fills a critical gap in the literature by providing data specific to Iraq, where comparative analyses of these scoring systems are lacking. Insights gained from this study could inform local protocols, enhance triage efficiency, and improve patient outcomes in Iraqi emergency departments .

ELIGIBILITY:
Inclusion Criteria:

* Patients with chest injuries that require clinical assessment using the Thorax Trauma Severity Score (TTSS) and the Trauma Injury Severity Score (TISS) within 6 hours of admission.
* Patients (or their legal guardians) must provide informed consent for participation in the study. This ensures ethical standards are maintained.
* Patients presenting with thoracic injuries, including rib fractures, pulmonary contusions, pneumothorax, hemothorax, and other chest-related injuries. This will include both isolated chest trauma and trauma with multiple injuries

Exclusion Criteria:

* Patients younger than 16 years.
* Patients with chest injuries caused by conditions unrelated to trauma, such as spontaneous pneumothorax, infections, or other medical conditions (e.g., non-traumatic rib fractures or cancer).
* Patients with severe co-morbidities (e.g., terminal illnesses, advanced stages of cancer, or end-stage organ failure) that would significantly affect outcomes unrelated to the chest trauma.
* Patients with pre-existing severe neurological conditions or other comorbidities that would interfere with trauma assessment and clinical management (e.g., severe brain injury, vegetative state).
* Patients or their legal representatives who refuse consent for participation in the study.
* Pregnant women due to potential risks associated with trauma and interventions during pregnancy.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of adult patients (18 years and older) who present to the Emergency Department (ER) of Al-Kadhimiya Teaching Hospital with chest trauma. This population will be classified based on the severity of their injuries, ranging from minor to critical, and include both blunt and penetrating trauma cases.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
In hospital mortality | In-Hospital Phase (average of 7-10 days through discharge)
  Mortality (death) during hospitalization.
Accuracy Assessment of Thorax Trauma Severity Score (TTSS) | the first 6 hours after ER admission
  Range: from 0 to 25, with higher scores indicating more severe thoracic trauma.
Accuracy Assessment of Trauma and Injury Severity Score (TRISS) | the first 6 hours after ER admission
  Range: 0 (represents a 0% probability of survival) to 1 (represents a 100% probability of survival), with higher scores indicating greater trauma severity.

SECONDARY OUTCOMES:
Length of Hospitalization | Up to discharge, an average of 7-10 days
  Description: The total duration of a patient's stay in the hospital, measured from the date of admission to the date of discharge. This includes all days spent in general wards, intensive care units (ICU), and other hospital departments as part of their treatment course.
Rate of admission to the intensive care unit (ICU) | Up to discharge, an average of 7-10 days
  The requirement for admission to the intensive care unit (ICU) is determined by the presence of severe clinical deterioration, significant complications, or the need for advanced monitoring and life-support measures.

CONTACTS AND LOCATIONS:
Overall Officials: Yaser aamer Eisa Alhaibi, Assistant professor, Study Director — College Of Medicine - Nahrain University
Locations (1):
- College of Medicine - Al-Nahrain University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Indurkar SK Sr, Ghormade PS, Akhade S, Sarma B. Use of the Trauma and Injury Severity Score (TRISS) as a Predictor of Patient Outcome in Cases of Trauma Presenting in the Trauma and Emergency Department of a Tertiary Care Institute. Cureus. 2023 Jun 14;15(6):e40410. doi: 10.7759/cureus.40410. eCollection 2023 Jun. PMID 37456404
- [Result] Zahran, M.R., Elwahab, A.A.E.M.A., El Nasr, M.M.A. et al. Evaluation of the predictive value of thorax trauma severity score (TTSS) in thoracic-traumatized patients. Cardiothorac Surg 28, 3 (2020). https://doi.org/10.1186/s43057-020-0015-7
- [Result] Imhoff BF, Thompson NJ, Hastings MA, Nazir N, Moncure M, Cannon CM. Rapid Emergency Medicine Score (REMS) in the trauma population: a retrospective study. BMJ Open. 2014 May 2;4(5):e004738. doi: 10.1136/bmjopen-2013-004738. PMID 24793256
- [Result] Karajizadeh M, Nasiri M, Yadollahi M, Zolfaghari AH, Pakdam A. Mortality Prediction from Hospital-Acquired Infections in Trauma Patients Using an Unbalanced Dataset. Healthc Inform Res. 2020 Oct;26(4):284-294. doi: 10.4258/hir.2020.26.4.284. Epub 2020 Oct 31. PMID 33190462
- [Result] Konesky KL, Guo WA. Revisiting traumatic cardiac arrest: should CPR be initiated? Eur J Trauma Emerg Surg. 2018 Dec;44(6):903-908. doi: 10.1007/s00068-017-0875-6. Epub 2017 Nov 25. PMID 29177620
- [Result] Mulvey HE, Haslam RD, Laytin AD, Diamond CA, Sims CA. Unplanned ICU Admission Is Associated With Worse Clinical Outcomes in Geriatric Trauma Patients. J Surg Res. 2020 Jan;245:13-21. doi: 10.1016/j.jss.2019.06.059. Epub 2019 Aug 5. PMID 31394403
- [Result] Todd KH, Lee T, Hoffman JR. The effect of ethnicity on physician estimates of pain severity in patients with isolated extremity trauma. JAMA. 1994 Mar 23-30;271(12):925-8. PMID 8120961
- [Result] Mondello S, Cantrell A, Italiano D, Fodale V, Mondello P, Ang D. Complications of trauma patients admitted to the ICU in level I academic trauma centers in the United States. Biomed Res Int. 2014;2014:473419. doi: 10.1155/2014/473419. Epub 2014 Jun 3. PMID 24995300
- [Result] Ramos-Pascua LR. Complications and trauma sequelae. Injury. 2018 Sep;49 Suppl 2:S1-S2. doi: 10.1016/j.injury.2018.06.045. Epub 2018 Jul 7. No abstract available. PMID 30097308
- [Result] Haagsma JA, Graetz N, Bolliger I, Naghavi M, Higashi H, Mullany EC, Abera SF, Abraham JP, Adofo K, Alsharif U, Ameh EA, Ammar W, Antonio CA, Barrero LH, Bekele T, Bose D, Brazinova A, Catala-Lopez F, Dandona L, Dandona R, Dargan PI, De Leo D, Degenhardt L, Derrett S, Dharmaratne SD, Driscoll TR, Duan L, Petrovich Ermakov S, Farzadfar F, Feigin VL, Franklin RC, Gabbe B, Gosselin RA, Hafezi-Nejad N, Hamadeh RR, Hijar M, Hu G, Jayaraman SP, Jiang G, Khader YS, Khan EA, Krishnaswami S, Kulkarni C, Lecky FE, Leung R, Lunevicius R, Lyons RA, Majdan M, Mason-Jones AJ, Matzopoulos R, Meaney PA, Mekonnen W, Miller TR, Mock CN, Norman RE, Orozco R, Polinder S, Pourmalek F, Rahimi-Movaghar V, Refaat A, Rojas-Rueda D, Roy N, Schwebel DC, Shaheen A, Shahraz S, Skirbekk V, Soreide K, Soshnikov S, Stein DJ, Sykes BL, Tabb KM, Temesgen AM, Tenkorang EY, Theadom AM, Tran BX, Vasankari TJ, Vavilala MS, Vlassov VV, Woldeyohannes SM, Yip P, Yonemoto N, Younis MZ, Yu C, Murray CJ, Vos T. The global burden of injury: incidence, mortality, disability-adjusted life years and time trends from the Global Burden of Disease study 2013. Inj Prev. 2016 Feb;22(1):3-18. doi: 10.1136/injuryprev-2015-041616. Epub 2015 Dec 3. PMID 26635210
- [Result] GBD 2021 Causes of Death Collaborators. Global burden of 288 causes of death and life expectancy decomposition in 204 countries and territories and 811 subnational locations, 1990-2021: a systematic analysis for the Global Burden of Disease Study 2021. Lancet. 2024 May 18;403(10440):2100-2132. doi: 10.1016/S0140-6736(24)00367-2. Epub 2024 Apr 3. PMID 38582094
- [Result] Lafta RK, Al-Nuaimi MA. National perspective on in-hospital emergency units in Iraq. Qatar Med J. 2013 Nov 1;2013(1):19-27. doi: 10.5339/qmj.2013.4. eCollection 2013. PMID 25003053
- [Result] Donaldson RI, Shanovich P, Shetty P, Clark E, Aziz S, Morton M, Hasoon T, Evans G. A survey of national physicians working in an active conflict zone: the challenges of emergency medical care in Iraq. Prehosp Disaster Med. 2012 Apr;27(2):153-61. doi: 10.1017/S1049023X12000519. Epub 2012 May 17. PMID 22591705